CLINICAL TRIAL: NCT07131605
Title: Effects of Bariatric Surgery on Cardiovascular Risk Profile in Relation to Inflammatory Parameters: Endothelial Phenotyping and Analysis of the Cross-talk Between Adipose Tissue and Endothelium
Acronym: BARIHEART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BARIHEART
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Obesity (Disorder)
Keywords: Obesity Cardiovascular risk, Metabolic impact, Bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Defecation; Urination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who are hospitalized and undergoing either gastric bypass or sleeve gastrectomy surgery (Other)
  Interventions: Other: Before bariatric surgery, both blood and biological samples (stool and urine) will be collected. Patients will also undergo a cardiology examination

INTERVENTIONS:
Other: Before bariatric surgery, both blood and biological samples (stool and urine) will be collected. Patients will also undergo a cardiology examination — This study includes a comprehensive set of laboratory and clinical investigations to evaluate the cardiovascular and metabolic impact of obesity and its modulation after bariatric surgery. Multiple biological samples (blood, urine, stool, and omental adipose tissue) will be collected at baseline and during follow-up.

SUMMARY:
This research project aims to study how obesity affects the heart and metabolism, and how these effects change after significant weight loss following bariatric surgery. In particular, we want to look at how blood vessels and fat tissue function in people with obesity, to detect early signs of vascular problems and understand how fat tissue communicates with blood vessels.

Our main idea is that obesity disrupts the normal function of blood vessels, partly due to substances released by fat tissue and changes in gut bacteria. We believe that 6 and 12 months after surgery - with proper weight loss - these problems will gradually improve. We expect to see better blood vessel function and lower levels of inflammation and fat-related substances in the blood, which could significantly reduce the overall risk of heart disease.

DETAILED DESCRIPTION:
The pathogenesis of obesity is multifactorial, involving dietary, socioeconomic, genetic, and metabolic factors. The accumulation of adipose tissue-especially abdominal fat-is only one aspect of the disease. Visceral fat, in fact, produces pro-inflammatory cytokines (adipocytokines) that contribute to the local recruitment of activated inflammatory macrophages (known as M1). These cells progressively accumulate in the adipose tissue and further amplify the inflammatory response.

Endothelial dysfunction, defined as the inability of the endothelium to regulate key vascular functions (such as vasodilation, coagulation, and permeability), is considered the earliest pathological event leading to atherosclerosis. In obesity, systemic inflammation, adipose tissue dysfunction, oxidative stress, and the presence of other risk factors contribute to impaired endothelial homeostasis-events that occur well before clinically evident cardiovascular (CV) disease.

Bariatric surgery has proven effective not only in reducing body weight but also in improving obesity-related comorbidities, particularly those involving the cardiovascular system. The hypothesis that weight loss also restores endothelial homeostasis-by interrupting the positive inflammatory feedback loop driven by fat accumulation-is supported by recent literature. However, the timing of functional recovery, as well as the influence of individual differences and cardiovascular risk factors on this process, remains unclear. Moreover, the mechanisms underlying adipose tissue-endothelium interactions are still only partially understood.This experimental project aims to study the cardiovascular and metabolic impact of obesity, and how this changes in response to the drastic weight loss induced by bariatric surgery.

Specifically, we plan to analyze endothelial homeostasis and adipose tissue dysfunction in these patients, in order to detect subclinical vascular alterations and explore potential mechanisms of cross-talk between adipocytes and the endothelium.

Our central hypothesis is that obesity leads to altered endothelial homeostasis, driven by mediators released from adipose tissue and by changes in the gut microbiota. We expect that, at 6 and 12 months after surgery-and with adequate weight loss-there will be progressive resolution of endothelial dysfunction, along with a reduction in circulating adipose-specific mediators and inflammatory markers, ultimately leading to a significant improvement in overall cardiovascular risk profile.

ELIGIBILITY:
Inclusion Criteria:

Adults (≥ 18 years old); Patients with obesity (Body Mass Index ≥ 30 kg/m²); Patients scheduled to undergo bariatric surgery via mini-gastric bypass or sleeve gastrectomy; Patients able to give their consent and to provide signed and dated informed consent for the processing of personal data; Willingness to attend follow-up visits and undergo all assessments required by the study protocol.

Exclusion Criteria:

Active systemic inflammatory diseases (e.g., chronic inflammatory bowel diseases, chronic rheumatologic diseases); Acute or chronic infections Severe anemia or coagulation disorders; Moderate to severe chronic kidney disease; Active malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2026-11-11 (Estimated)

PRIMARY OUTCOMES:
changes at the vascular tissue | 12 months
  Measurement of circulating endothelial cells ( cells/µL)
To analyze the changes adipose tissue | from enrollment to the end of study at 12 month
  Cardiac CT for assessment of epicardial adipose tissue. Volume quantification by tracing (cm³)

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared. However, de-identified data may be made available to qualified researchers upon reasonable request to the study center and the Principal Investigator. All data will be processed in compliance with the General Data Protection Regulation (GDPR - EU Regulation 2016/679), ensuring the confidentiality, integrity, and protection of participants' personal information."